CLINICAL TRIAL: NCT06289530
Title: A Multicenter Prospective Cohort Study on the Association Between Perioperative Blood and Interstitial Fluid Glucose Level and Clinically Relevant Postoperative Pancreatic Fistula in Different Pancreatic Surgeries
Brief Title: Association Between Perioperative Blood and Interstitial Fluid Glucose Level and Clinically Relevant Postoperative Pancreatic Fistula in Different Pancreatic Surgeries
Acronym: CR-POPF
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2023XAGG0070-1
Record Dates: First submitted 2024-02-25; First posted 2024-03-04 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-03

CONDITIONS: Postoperative Pancreatic Fistula
Keywords: clinically relevant postoperative pancreatic fistula; pancreatic surgery; perioperative interstitial fluid glucose level

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This observational study was conducted in patients undergoing elective pancreaticoduodenectomy or distal pancreatectomy. It mainly answers the following two main questions:

1. What are the risk factors for clinically relevant postoperative pancreatic fistula in different pancreatic surgeries?
2. What is the correlation between perioperative blood and interstitial fluid glucose level and clinically relevant postoperative pancreatic fistula in different pancreatic surgeries？

Participants were not required to perform additional research work other than the usual postoperative follow-up within 30 days after surgery. No control group was set in this study, and no additional clinical intervention was performed.

DETAILED DESCRIPTION:
CR-POPF is a multi-center observational prospective cohort study. The research team focuses on whether perioperative abnormal hyperglycemia can independently predict the occurrence of CR-POPF. It is proposed to realize the dynamic monitoring of perioperative blood glucose level by non-invasive continuous glucose monitoring (CGM), and perioperative continuous glucose monitoring can reflect the overall blood glucose trend and mode, which is helpful to further explore the correlation between perioperative abnormal blood glucose level and CR-POPF.

The investigators expect to enroll 600 patients. Based on our previous clinical experience, the incidence of postoperative pancreatic fistula is approximately 20%. We planned to enroll 600 patients during the 6-month enrollment period in three participating hospitals. The sample size would have a statistical power of 81.3% to detect an odds ratio (OR) greater than 1.34 or less than 0.75.

Measurement data consistent with normal distribution were expressed as mean ± standard deviation, and t-test was used for comparison between groups. When not consistent with normal distribution, the measurement data were expressed as quartiles, and the Wilcoxon-Mann-Whitney rank sum test was used for comparison between groups. Count data were expressed as frequency and percentage. Pearson chi-square test or Fisher's exact test was used for comparison between groups. The binary logistic regression method was used to screen the risk factors and stratify the risk levels, P < 0.05 was considered statistically significant. A generalized estimation equation model was constructed to analyze the correlation between continuous blood glucose monitoring values and postoperative pancreatic fistula. The dependent variable in the model is whether there is pancreatic fistula after operation. The dependent variable in the model was the presence or absence of postoperative pancreatic fistula, and the main variable was the continuous glucose monitoring (CGM) value. The connection function uses the binomial distribution logit function. The multiple measurements of the same patient are set as the group-level variable, and the autocorrelation matrix is selected according to the Quasi-likelihood under Independence Model Criterion (QIC) value of the model. In addition to analysis using generalized estimating equations, continuous glucose monitoring data will be constructed, such as an analysis of the association between pancreatic fistula and the area under the curve for measurement and time beyond normal glucose values. The statistical software was STATA ( version 15.0; stata Corp., Texas, USA ) and R 3.6.1 software ( R Foundation for Statistical Computing, Vienna, Austria ), bilateral P < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective pancreaticoduodenectomy
* Patients scheduled for distal pancreatectomy
* Patients scheduled for duodenum-preserving resection of pancreatic head.

Exclusion Criteria:

* Patients with functional pancreatic neuroendocrine tumors.
* Patients with previous pancreatic surgery.
* Patients with severe pancreatitis.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing elective pancreaticoduodenectomy or distal pancreatectomy from March 2024 to October 2024.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Clinically relevant postoperative pancreatic fistula | 30 days after surgery
  Clinically relevant postoperative pancreatic fistula is now redefined as a drain output of any measurable volume of fluid with an amylase level >3 times the upper limit of institutional normal serum amylase activity, associated with a clinically relevant development/condition related directly to the postoperative pancreatic fistula.

SECONDARY OUTCOMES:
Bile leakage | 30 days after surgery
  Bile leakage was defined as bilirubin concentration in the drain fluid at least 3 times the serum bilirubin concentration on or after postoperative day 3 or as the need for radiologic or operative intervention resulting from biliary collections or bile peritonitis.
Chyle leak | 30 days after surgery
  Chyle leak was defined as output of milky-colored fluid from a drain, drain site, or wound on or after postoperative day 3, with a triglyceride content greater than or equal to 110 mg/dL (1.2 mmol/L).
Postpancreatectomy hemorrhage | 30 days after surgery
  Postpancreatectomy hemorrhage is defined by 3 parameters: onset, location, and severity. The onset is either early (24 hours after the end of the index operation) or late (24 hours). The location is either intraluminal or extraluminal. The severity of bleeding may be either mild or severe.
Abdominal infection | 30 days after surgery
  Abdominal infection was defined as a patient with symptoms such as shivering, high fever, abdominal distension, intestinal paralysis and other symptoms 3 or more days after surgery lasting for more than 24 hours.Laboratory examination results showed significant increases in white blood cell count, procalcitonin, and hypersensitive C-reactive protein, and imaging examination showed accumulation of fluid in the abdominal cavity. The diagnosis can be confirmed by the detection of bacteria or fungi in abdominal drainage or paracentesis fluid.
Delayed gastric emptying | 30 days after surgery
  Delayed gastric emptying was defined as indwelling gastric tube for more than 3 days after surgery, or re-indwelling gastric tube after 3 days due to vomiting or abdominal distension, or still unable to tolerate solid food 7 days after surgery under the premise of unobstructed gastrointestinal or duodenojejunal anastomosis and no obstruction of the small intestine.

CONTACTS AND LOCATIONS:
Overall Officials: YuGuang Huang, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital,Chinese Academy of Medical Science and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lan L, Zhang Y, Zhang L, Zhang Y, Shen L, Huang Y. Association between perioperative continuous glucose monitoring and clinically relevant postoperative pancreatic fistula (CR-POPF) in pancreatic surgery: a protocol for a prospective cohort study. BMJ Open. 2025 Jun 17;15(6):e092046. doi: 10.1136/bmjopen-2024-092046. PMID 40527571